CLINICAL TRIAL: NCT00609999
Title: Phase I Study of Dasatinib Plus Erlotinib in Recurrent Malignant Glioma
Brief Title: Ph I Dasatinib + Erlotinib in Recurrent MG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002272
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2012-04

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; GBM; Recurrent MG; Erlotinib; Dasatinib; Brain tumor; Malignant glioma; Tarceva; Sprycel
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma | interventions — Erlotinib Hydrochloride; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum A (Experimental): Pts not on EIAEDs
  Interventions: Drug: Erlotinib and Dasatinib
- Stratum B (Experimental): Pts on EIAEDs
  Interventions: Drug: Erlotinib and Dasatinib

INTERVENTIONS:
Drug: Erlotinib and Dasatinib — You will begin study drug regimen on day 1 of cycle 1 w Dasatinib. If you are undergoing Dasatinib pharmacokinetic blood analysis, Dasatinib will be taken alone until initial PK assessments are collected. Erlotinib will be begin after initial Dasatinib PK assessments are collected & will continue to be administered w Dasatinib on continuous daily dosing schedule. Initial Dasatinib PK assessments will be collected over 24hrs between days 3-7 of cycle 1 & at end of cycle 1. If you are not undergoing Dasatinib PK collections you will begin both Dasatinib & Erlotinib together on day 1 of cycle 1. Both drugs will be given in continuous daily oral manner. Cycle is defined as Dasatinib & Erlotinib given daily for 28 days for purpose of scheduling evaluations.
  Other Names: Dasatinib; Erlotinib; Tarceva; Sprycel

SUMMARY:
Primary:

To determine maximum tolerated dose & dose limiting toxicity of dasatinib when combined w erlotinib among pts w recurrent MG

Secondary:

To further evaluate safety & tolerability of dasatinib + erlotinib To evaluate pharmacokinetics of dasatinib when administered w erlotinib among recurrent MG pts who are on & not on CYP-3A enzyme inducing anti-epileptic drugs To evaluate for anti-tumor activity with this regimen in this patient population

DETAILED DESCRIPTION:
Tarceva administered on continuous oral dosing schedule at 150 mg/day for pts not on EIAEDs & 450 mg/day for pts on EIAEDs. Starting dose level of dasatinib will be 100 mg once day via continuous oral daily dosing. Dasatinib will be increased in successive cohorts of enrolled pts. Pts will remain on treatment until excessive toxicity, progressive disease, withdrawal of consent/death.

Pts have confirmed diagnosis of recurrent/progressive WHO gr IV MG / WHO grade III MG. Phase I 3+3 dose escalation design w 2 independently escalated stratum: stratum A-pts not on CYP3A-enzyme inducing anti-epileptic drugs; stratum B-pts on EIAEDs. Assessment of safety will be based mainly on frequency of adverse events, particularly adverse events leading to discontinuation of treatment & on number of significant lab abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent/progressive WHO grade IV MG or WHO grade III MG. Pts with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO grade III / IV MG
* >18 yrs
* Karnofsky Performance Status >70 percent
* Pts presenting in 1st, 2nd / 3rd relapse. Prior therapy must have included external beam XRT
* Adequate bone marrow, liver & renal function as assessed by following:
* Hemoglobin>9.0g/dl
* ANC>1,500/mm3
* Platelet count>100,000/mm3
* Total bilirubin<1.5 x ULN
* ALT & AST<2.5 x ULN
* INR<1.5 or PT/PTT within normal limits. Pts receiving anti-coagulation treatment w low-molecular weight heparin allowed to participate, oral warfarin is not permitted
* Creatinine<1.5 x ULN
* Serum Na, K+, Mg2+, Phosphate & Ca2+ >LLN
* Interval<2 wks between prior surgical resection & initiation of study regimen
* Interval <12 weeks from completion of standard, daily XRT, unless one of following occurs: new area of enhancement on MRI imaging that is outside XRT field; biopsy proven recurrent tumor; / radiographic evidence of progressive tumor on 2 consecutive scans >4 wks apart.
* Interval <4weeks from prior chemotherapy unless there is unequivocal evidence of tumor progression & pt has recovered from all anticipated toxicities from prior therapy
* Interval <4weeks from prior investigational agent unless there is unequivocal evidence of tumor progression & pt has recovered from all anticipated toxicities from prior therapy
* Signed written informed consent including HIPAA according to institutional guidelines. Signed informed consent must be obtained prior to any study specific procedures
* If sexually active, pts will take contraceptive measures for duration of treatments & for 4 weeks following discontinuation of dasatinib & Erlotinib.
* Women of childbearing potential must have negative serum or urine pregnancy test within 72 hrs prior to start of study drug administration

Exclusion Criteria:

* No prior dasatinib / oral EGFR-inhibitor therapy
* Pregnancy/breast feeding
* History of significant concurrent illness

  ->3 prior episodes of progressive disease
* Significant cardiac disease
* Excessive risk of bleeding as defined by stroke <6 months, history of CNS / intraocular bleed,/ septic endocarditis.
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in study including any of following: pleural / pericardial effusion of any grade; uncontrolled diabetes; uncontrolled hypertension; active clinically serious infection >CTCAEv3 Gr2 requiring active intervention; history of clinically-significant bleeding diathesis or coagulopathy including platelet function disorder or acquired bleeding disorder within 1yr; impairment of GI function /GI disease that may significantly alter absorption of study regimen; ongoing or recent significant gastrointestinal bleeding
* Thrombolic or embolic events such as cerebrovascular accident including transient ischemic attacks <6 months
* Any hemorrhage/bleeding event >CTCAEv3AE Gr3 within 4wks of 1st dose of study drug
* Serious non-healing wound, ulcer, /bone fracture
* Major surgery, open biopsy /significant traumatic injury <4 weeks of 1st study drug
* Known HIV infection/chronic Hepatitis B/C
* Pt is <3yrs free of another primary malignancy except: if other primary malignancy is either not currently clinically significant/does not require active intervention. Existence of any other malignant disease is not allowed.
* Pts unwilling to/unable to comply with protocol including ability to swallow whole pills/presence of any malabsorption syndrome
* Concurrent administration of warfarin, rifampin/St. John's Wort
* Subjects w hypokalemia/hypomagnesemia if it cannot be corrected
* Prisoners/subjects who are compulsorily detained for treatment of either psychiatric/physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine MTD & DLT of Dasatinib when combined w Erlotinib among pts w Recurrent MG | 12 months

SECONDARY OUTCOMES:
To further evaluate safety & tolerability of Dasatinib + Erlotinib | 12 months
To evaluate the PK of Dasatinib when administered w Erlotinib among Recurrent MG pts who are on & not on EIAEDs | 12 months
To evaluate for anti-tumor activity w this regimen in this pt population | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/